CLINICAL TRIAL: NCT02570841
Title: Heat-, Cold-, and Mechanical Pain Thresholds Under Exposition of High Dose Topical Capsaicin
Brief Title: Pain Thresholds Under High-dose Topical Capsaicin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Astellas Pharma GmbH (Industry)
Responsible Party: Principal Investigator, E. Knolle, MD, Ao.Univ.-Prof. Dr. Erich Knolle, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FA738B0401
Record Dates: First submitted 2015-09-08; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: Heat pain threshold; Cold pain threshold; Mechanical pain threshold; High dose Capsaicin
MeSH Terms: conditions — Pain | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsaicin (Active Comparator): Treatment with Topical High dose Capsaicin
  Interventions: Drug: Topical High dose Capsaicin
- Placebo (Placebo Comparator): Treatment with Topical Placebo
  Interventions: Drug: Topical Placebo

INTERVENTIONS:
Drug: Topical High dose Capsaicin — Topical High dose Capsaicin exposure within an area of 3x3 cm for 60 minutes
  Other Names: Topical Capsaicin 8%; Qutenza® patch
  Arms: Capsaicin
Drug: Topical Placebo — Placebo exposure within an area of 3x3 cm for 60 minutes
  Other Names: Demo patch
  Arms: Placebo

SUMMARY:
Aim of the study is to determine heat pain thresholds (HPT in °C) and cold pain thresholds (CPT in °C) during topical capsaicin 8% application, and mechanical pain thresholds (MPT in g) immediately after to find out the exact skin temperature by which capsaicin initiates the application pain (heat pain threshold, HPT in °C) but also the temperature by which capsaicin does not yet trigger a cold pain (cold pain threshold, CPT in °C). Moreover the investigators want to find out the mechanical pain threshold in g from topical capsaicin and to verify a prolonged effect of capsaicin on the pain thresholds.

DETAILED DESCRIPTION:
Capsaicin is the main pungent ingredient in chili peppers. Topical capsaicin 8% is used for the treatment of peripheral neuropathic pain. Application of capsaicin 8% provokes distinct pain by activating the transient receptor potential vanilloid 1 (TRPV1) receptor. Cooling the skin results in a reliable prevention of the application pain. However, the necessary cooling temperature and if cooling itself produces application pain, is unknown.

Materials and Methods: 10 female and 10 male healthy volunteers will be enrolled in a randomised, double blind, placebo controlled, cross-over study. The left or right forearm of each subject is going to be treated with a capsaicin 8% patch (QUTENZA, Astellas Pharma, Tokyo, Japan) of 9 cm² or a placebo patch (Demo patch, Astellas Pharma, Tokyo, Japan) of the same size for 60 min. Then the other forearm (which has not been tested before) will be treated with the remaining patch. During capsaicin and placebo exposure HPT in °C and CPT in °C are going to be obtained by the thermode of a thermal sensory analyser, TSA-II (Medoc Ltd., Ramat Yishai, Israel). Temperature increase/decrease of the thermode will be stopped, as soon as the subject presses a switch because of a beginning pain sensation. Immediately after exposure a pin prick test will be performed 5 times in a row by pressing a Mini-Spike (B. Braun Melsungen AG, Melsungen, Germany) slowly against the skin of the application areal to determine the pressure necessary to provoke a sharp pain (Mechanical pain threshold in g). 2 weeks later HPT, CPT, and MPT will be determined again in the areas of capsaicin and placebo exhibition.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers 18 ore more years old

Exclusion Criteria:

* dermatologic or neurologic injuries on both thighs, (possible) pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Heat pain threshold (HPT) in degrees Celsius (°C) | 60 minutes during topical highdose Capsaicin/Placebo exposure
  During capsaicin and placebo exposure HPT in degrees Celsius (°C) is determined by a thermal sensory analyser TSA-II (Medoc Ltd.)

SECONDARY OUTCOMES:
Cold pain threshold (CPT) in degrees Celsius (°C) | 60 minutes during topical highdose Capsaicin/Placebo exposure
  During capsaicin and placebo exposure CPT in degrees Celsius (°C) is determined by a thermal sensory analyser TSA-II (Medoc Ltd.)
Mechanical pain threshold (MPT) in grams (g) | Immediately after topical highdose Capsaicin/Placebo exposure
  After capsaicin and placebo exposure MPT in grams (g) is determined by pressing a Mini-Spike (B. Braun Melsungen AG, Melsungen, Germany) slowly against the skin of the application areal to determine the pressure necessary to provoke a sharp pain
HPT in degrees Celsius (°C) | 2 weeks after exposure
  HPT in degrees Celsius (°C) will be determined again in the areas of capsaicin and placebo Exhibition
CPT in degrees Celsius (°C) | 2 weeks after exposure
  CPT in degrees Celsius (°C) will be determined again in the areas of capsaicin and placebo Exhibition
MPT in grams (g) | 2 weeks after exposure
  MPT in grams (g) will be determined again in the areas of capsaicin and placebo Exhibition

CONTACTS AND LOCATIONS:
Overall Officials: Erich Knolle, MD, Principal Investigator — Department of Anesthesia, Critical Care and Pain Medicine
Locations (1):
- Department of Anesthesia, Critical Care and Pain Medicine, Vienna, Vienna, Austria